CLINICAL TRIAL: NCT04761887
Title: Pilot Study on the Thermal Effects of Local Anesthetics
Brief Title: Cool Pre-operative TAP Blocks
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment (insufficient funds and reduced access to patients related to COVID protocols)
Sponsor: Daniel Wambold (Other)
Responsible Party: Sponsor-Investigator, Daniel Wambold, Study Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 57733
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Anesthetics, Local
Keywords: ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cool Block (Experimental): Ropivacaine administered at approximately 4C, via a TAP block.
  Interventions: Drug: Cool Ropivacaine Block
- Room Temp Block (Active Comparator): Ropivacaine administered at approximately 20-25C, via a TAP block.
  Interventions: Drug: Room Temp Ropivacaine Block

INTERVENTIONS:
Drug: Cool Ropivacaine Block — Ropivacaine is cooled.
  Arms: Cool Block
Drug: Room Temp Ropivacaine Block — Room Temp Block
  Arms: Room Temp Block

SUMMARY:
This is a pilot study of approximately 20 pre-operative patients scheduled for a transversus abdominis plane (TAP) block as pain management for a previously scheduled surgery. Subjects will be randomly assigned to receive either cooled ropivacaine (4°C) during a TAP block or room temperature (between 20-25°C) ropivacaine during the block. The effects of a TAP block generally diminish within 24 hours. We believe that cooling ropivacaine before administration may slightly prolong the analgesic effects of the block and delay time before additional analgesic is requested, resulting in less opioid use following surgery.

DETAILED DESCRIPTION:
After consenting, subjects will be randomized to receive either cooled ropivacaine, administered at approximately 4°C) or room temperature ropivacaine, administered at approximately 20-25°C), during an ultrasound-guided TAP block. Time to anesthesia, or loss of sensation, will be recorded for each subject by a single evaluator, employing the pinch technique and thermosensory perception, using a glove, filled with a slurry of ice water placed on both anesthetized and non-anesthetized areas, for approximately 5 seconds. Time to anesthesia will be recorded when there is a definitive difference on a categorical scale (painful/not painful or cold/not cold) as measured by the subject, between the anesthetized and non-anesthetized areas. Safety outcomes and opioid morphine equivalency will be recorded for all subjects, for approximately 48 hours following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, aged =18 years of age.
2. Patients, scheduled for surgery, with an order for a TAP block.

Exclusion Criteria:

1. Patients with a history of opioid use disorder.
2. Patients, which are scheduled as the first case of the day.
3. Patients with any history of paralysis/palsy.
4. Patients with a history of sensitivity to local anesthetics, including ropivacaine.
5. Patients, whose blocks are scheduled to be administered by a PGY-1 or PGY-2 resident.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Time to block of pain and thermosensory perception | 35 minutes

SECONDARY OUTCOMES:
Morphine equivalency units of adjunct pain medications | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wambold, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No